CLINICAL TRIAL: NCT02746198
Title: A Randomized Double-blind Placebo-controlled Clinical Pilot Trial on the Effect of a Probiotic Fermented Drink on Antibiotic-associated Diarrhea (AAD) in Patients With Helicobacter Pylori Eradication Therapy
Brief Title: Clinical Pilot Trial on the Effect of a Probiotic Fermented Drink on Antibiotic-associated Diarrhea (AAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Research Center Kiel GmbH (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14DE-KIEL-HPAAD1
Record Dates: First submitted 2016-04-12; First posted 2016-04-21 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Antibiotic-associated Diarrhea
Keywords: Probiotics, Antibiotics, AAD, Helicobacter p.
MeSH Terms: interventions — calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Verum (Experimental): 2 bottles (á 65ml) of a probiotic dairy drink consumed daily for 6 weeks
  Interventions: Other: probiotic dairy drink
- Placebo (Placebo Comparator): 2 bottles (á 65ml) of a dairy drink containing chemically acidified milk without bacterial strains consumed daily for 6 weeks
  Interventions: Other: acidified milk

INTERVENTIONS:
Other: probiotic dairy drink
  Other Names: verum
  Arms: Verum
Other: acidified milk
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to estimate the effect of a probiotic dairy drink on occurrence and duration of AAD and gastrointestinal symptoms during Helicobacter pylori (Hp) eradication therapy and during 4 weeks thereafter and calculating the sample size for a confirmatory study.

DETAILED DESCRIPTION:
Helicobacter p. positive subjects aged ≥18 years with an indication for Helicobacter pylori (Hp) eradication recommended by a gastroenterologist should be included in the study. Subjects should be willing to consume 2 servings of the study product per day for 6 weeks, and to undergo an Hp eradication therapy for 14 days starting with the consumption period.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, both genders, aged ≥ 18 y
* Helicobacter p. infected individuals, to which eradication therapy has been recommended by gastroenterologists
* Willingness to undergo the Helicobacter p. eradication therapy
* Willingness to abstain from food and supplements containing probiotics, prebiotics and fermented products except the study product
* Written informed consent

Exclusion Criteria:

* Subjects currently enrolled in another interventional trial
* subjects having finished another interventional trial within the last 4 weeks before inclusion
* incapacity to comply with the study protocol
* allergy or hypersensitivity to any component of the test product (allergy against milk protein)
* allergy or hypersensitivity to any component of the eradication therapy (e.g. penicillin allergy)
* acute GIT infections
* chronic inflammatory bowel diseases (IBD)
* irritable bowel syndrome (IBS)
* any episode of diarrhea according to WHO criteria during the last 4 weeks before inclusion
* history of lactose intolerance
* severe chronic disease (cancer, malabsorption, malnutrition, severe chronic inflammatory diseases (except chronic gastritis), renal, hepatic or cardiac diseases, artificial cardiac valve, COPD, respiratory insufficiency)
* history of active or persistent hepatitis B and C
* known congenital, acquired or iatrogenic immunodeficiency (e.g. HIV, chemotherapy, immunosuppression)
* systemic treatment with antibiotics during the last 4 weeks before inclusion
* systemic treatment likely influencing absorption, metabolism and excretion of food ingredients (metoclopramide, laxatives, body weight management and/or medication etc.)
* systemic treatment likely interfering or influencing effectiveness of the eradication drugs used e.g. ergotamine, statins, clopidogrel
* regular medical treatment including OTC, which may have impact on the study aims (e.g. probiotics, antibiotic drugs, laxatives etc.)
* severe neurological, cognitive or psychiatric diseases
* surgery or intervention requiring general anaesthesia within 2 months before the study
* vegan
* eating disorders (e.g. anorexia, bulimia)
* present alcohol and drug abuse
* pregnancy or lactation
* legal incapacity
* blood parameters:

  * Hb < 12 g/dL
  * liver transaminases (ALT, AST) > 2-fold increased
  * serum creatinine out of the normal range
* subjects who are scheduled to undergo hospitalization during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of antibiotic-associated diarrhea (AAD) | 6 weeks
  Occurrence of antibiotic-associated diarrhea (AAD) (as defined by number of subjects with diarrhea within the intervention period of 6 weeks after starting antibiotic treatment; diarrhea is defined according WHO

SECONDARY OUTCOMES:
Cumulated duration of antibiotic-associated diarrhea (AAD) | 6 weeks
  Number of days with diarrhea within the intervention period
Gastrointestinal Symptom Rating Scale | 6 weeks
  Standardized questionnaire according Dimenäs et al.
Cumulative sverity of antibiotic-associated diarrhea (AAD) | 6 weeks
  Sum of the values (obtained by transformation of Bristol stool form types) of all stools during days with diarrhea (transformation of Bristol scale types is defined: type 1 to 4 = 0; type 5 = 1; type 6 = 2 and type 7 = 3)

CONTACTS AND LOCATIONS:
Overall Officials: Chiyuki Kajita, Study Chair — Yakult Europe BV
Locations (1):
- CRC Clinical Research Center Kiel, Kiel, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No